CLINICAL TRIAL: NCT02763319
Title: A Phase 2/3, Randomised, Multicentre Study of Tafasitamab With Bendamustine Versus Rituximab With Bendamustine in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (R-R DLBCL) Who Are Not Eligible for High-Dose Chemotherapy (HDC) and Autologous Stem-Cell Transplantation (ASCT)
Brief Title: A Trial to Evaluate the Efficacy and Safety of Tafasitamab With Bendamustine (BEN) Versus Rituximab (RTX) With BEN in Adult Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Acronym: B-MIND
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOR208C204; 2014-004689-11 (EudraCT Number)
Record Dates: First submitted 2016-04-30; First posted 2016-05-05 (Estimated); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse Large B-cell Lymphoma; bendamustine; rituximab; combination therapy; CD19 monoclonal antibody; transplant ineligible
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; tafasitamab; Bendamustine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor: blinding on treatment group
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tafasitamab and bendamustine (Experimental): Tafasitamab and bendamustine
  Interventions: Drug: Tafasitamab; Drug: Bendamustine (BEN)
- Rituximab and bendamustine (Active Comparator): Rituximab and bendamustine
  Interventions: Drug: Rituximab (RTX); Drug: Bendamustine (BEN)

INTERVENTIONS:
Drug: Rituximab (RTX) — Rituximab: Dose: 375 mg/m2 IV
  Other Names: Rituxan; Mab Thera
  Arms: Rituximab and bendamustine
Drug: Tafasitamab — Tafasitamab: Tafasitamab dose: 12 mg/kg intravenously (IV)
  Arms: Tafasitamab and bendamustine
Drug: Bendamustine (BEN)
  Other Names: Levact/Treanda

SUMMARY:
The purpose of the study is to compare the safety and efficacy of Tafasitamab with BEN versus RTX with BEN in adult patients with relapsed of refractory DLBCL.

DETAILED DESCRIPTION:
This is a randomised, two-arm, multicentre, open-label phase II/III efficacy and safety study of Tafasitamab in combination with BEN versus RTX in combination with BEN given to adult patients who have relapsed after or are refractory to at least one but no more than three prior systemic therapies and have failed, or are not candidates for HDC and ASCT, and have thus exhausted their therapeutic options of demonstrated clinical benefit. At least one prior therapy line must have included a CD20-targeted therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age ≥18 years
2. Histologically confirmed diagnosis, according to the World Health Organization (WHO, 2008) classification, of: DLBCL NOS, THRLBCL, EBV-positive DLBCL, composite lymphoma with a DLBCL component with a DLBCL relapse subsequent to DLBCL treatment, disease transformed from an earlier diagnosis of low grade lymphoma (i.e. an indolent pathology such as follicular lymphoma, marginal zone lymphoma) into DLBCL with a DLBCL relapse subsequent to DLBCL treatment.
3. Fresh tumour tissue for central pathology review must be provided as an adjunct to participation in this study. Should it not be possible to obtain a fresh tumour tissue sample, archival paraffin embedded tumour tissue acquired ≤3 years prior to screening for this protocol must be available for this purpose.
4. Patients must have:

   1. relapsed or refractory DLBCL
   2. at least one bidimensionally measurable disease site. The lesion must have a greatest transverse diameter of ≥1.5 cm and greatest perpendicular diameter of ≥1.0 cm at baseline. The lesion must be positive on PET scan
   3. received at least one, but no more than three previous systemic therapy lines for the treatment of DLBCL. At least one previous therapy line must have included a CD20-targeted.
   4. ECOG 0 to 2
5. Patients after failure of ASCT or patients considered in the opinion of the investigator currently not eligible for HDC with subsequent ASCT.
6. Patients must meet the following laboratory criteria at Screening:

   1. ANC ≥1.5 × 109/L (unless secondary to bone marrow involvement by DLBCL)
   2. PLTs ≥90 × 109/L (unless secondary to bone marrow involvement by DLBCL) and absence of active bleeding
   3. total serum bilirubin ≤2.5 × ULN unless secondary to Gilbert's syndrome (or pattern consistent with Gilbert's) or documented liver involvement by lymphoma. Patients with Gilbert's syndrome or documented liver involvement by lymphoma may be included if their total bilirubin is ≤5 x ULN
   4. ALT, AST and AP ≤3 × ULN or <5 × ULN in cases of documented liver involvement by lymphoma
   5. serum creatinine ≤2.0 x ULN or creatinine clearance must be ≥40 mL/min calculated using a standard Cockcroft-Gault formula (Cockroft & Gault, 1976)
7. For a female of childbearing potential (FCBP), a negative pregnancy test must be confirmed before enrolment. An FCBP must commit to take highly effective contraceptive precautions without interruption during the study and for 3, 6 or 12 months after the last dose of Tafasitamab, BEN or RTX respectively, whichever is later. An FCBP must refrain from breastfeeding and donating blood or oocytes during the course of the study and for 3, 6 or 12 months after the last dose of Tafasitamab, BEN or RTX respectively, whichever is later. Restrictions concerning blood donations apply as well to females who are not of childbearing potential.
8. Males must use an effective barrier method of contraception without interruption during the study and for 3, 6 or 12 months after the last dose of Tafasitamab, BEN or RTX respectively, whichever is later, if the patient is sexually active with an FCBP. Males must refrain from donating blood or sperm during study participation and for 3, 6 or 12 months after the last dose of Tafasitamab, BEN or RTX respectively, whichever is later.
9. In the opinion of the investigator, the patients must:

   1. be able to comply with all study-related procedures, medication use, and evaluations
   2. be able to understand and give informed consent
   3. not be considered to be potentially unreliable and/or not cooperative.

EXCLUSION CRITERIA:

1. Patients who have: any other histological type of lymphoma including, e.g., primary mediastinal (thymic) large B-cell lymphoma (PMBL) or Burkitt's lymphoma, primary refractory DLBCL, patients with known "double/triple hit" DLBCL genetics, CNS lymphoma involvement in present or past medical history
2. Patients who had a major surgery less than 30 days prior to Day 1 dosing
3. Patients who have, within 14 days prior to Day 1 dosing:

   1. not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma-specific therapy
   2. received live vaccines
   3. required parenteral antimicrobial therapy for active, intercurrent systemic infections
4. Patients who:

   1. in the opinion of the investigator, have not recovered sufficiently from the adverse toxic effects of prior therapies, major surgeries or significant traumatic injuries
   2. were previously treated with CD19-targeted therapy or BEN
   3. have a history of previous severe allergic reactions to compounds of similar biological or chemical composition to Tafasitamab, RTX, murine proteins or BEN, or the excipients contained in the study drug formulations
   4. have undergone ASCT within a period of ≤3 months prior to signing the informed consent form. Patients who have a more distant history of ASCT must exhibit full haematological recovery before enrolment into the study.
   5. have undergone previous allogeneic stem cell transplantation
   6. concurrently use other anticancer or experimental treatments
5. Prior history of malignancies other than DLBCL, unless the patient has been free of the disease for ≥3 years prior to Screening. Exceptions to the ≥3-year time limit include history of the following:

   1. basal cell carcinoma of the skin
   2. squamous cell carcinoma of the skin
   3. carcinoma in situ of the cervix, breast and bladder

   f) incidental histological finding of prostate cancer (Tumour/Node/Metastasis [TNM] stage of T1a or T1b)
6. Patients with:

   1. positive hepatitis B and/or C serology
   2. known seropositivity for or history of active viral infection with HIV
   3. evidence of active, severe uncontrolled systemic infections or sepsis
   4. a history or evidence of severely immunocompromised state
   5. a history or evidence of severe hepatic impairment (total serum bilirubin > 3 mg/dL), jaundice unless secondary to Gilbert's syndrome or documented liver involvement by lymphoma
   6. a history or evidence of clinically significant cardiovascular, cerebrovascular, CNS and/or other disease that, in the investigator's opinion, would preclude participation in the study or compromise the patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Director, Study Director — Incyte Corporation
Locations (141):
- United States (18):
  - MorphoSys Research Site, Anaheim, California
  - MorphoSys Research Site, Bakersfield, California
  - Morphosys Research Site, Burbank, California
  - Morphosys Research Site, Fresno, California
  - MorphoSys Research Site, Los Angeles, California
  - MorphoSys Research Site, Whittier, California
  - MorphoSys Research Site, Plainville, Connecticut
  - MorphoSys Research Site, Skokie, Illinois
  - MorphoSys Research Site, Detroit, Michigan
  - MorphoSys Research Site, Rochester, Minnesota
  - MorphoSys Research Site, Hattiesburg, Mississippi
  - Morphosys Research site, Jackson, Mississippi
  - Morphosys Research Site, Morristown, New Jersey
  - MorphoSys Research Site, New York, New York
  - MorphoSys Research Site, Stony Brook, New York
  - MorphoSys Research Site, Oklahoma City, Oklahoma
  - MorphoSys Research Site, Knoxville, Tennessee
  - Morphosys Research Site, Lubbock, Texas
- Australia (12):
  - MorphoSys Research Site, Adelaide
  - MorphoSys Research Site, Albury
  - MorphoSys Research Site, Bedford Park
  - MorphoSys Research Site, Box Hill
  - MorphoSys Research Site, Concord
  - MorphoSys Research Site, Frankston
  - MorphoSys Research SIte, Garran
  - MorphoSys Research Site, Geelong
  - MorphoSys Research Site, Gosford
  - MorphoSys Research Site, Nedlands
  - MorphoSys Research Site, South Brisbane
  - MorphoSys Research Site, St Albans
- MorphoSys Research Site, Innsbruck, Austria
- Canada (8):
  - Morphosys Research Site, Edmonton, Alberta
  - MorphoSys Research Site, Winnipeg, Manitoba
  - MorphoSys Research Site, Saint John, New Brunswick
  - Morphosys Research Site, St. John's, Newfoundland and Labrador
  - MorphoSys Research Site, Kingston, Ontario
  - MorphoSys Research Site, Greenfield Park, Quebec
  - Morphosys Research Site, Montreal, Quebec
  - MorphoSys Research Site, Saskatoon
- MorphoSys Research Site, Zagreb, Croatia
- Czechia (4):
  - MorphoSys Research Site, Hradec Králové
  - Morphosys Research site, Olomouc
  - Morphosys Research Site, Prague
  - MorphoSys Research Site, Prague
- Finland (2):
  - MorphoSys Research Site, Oulu
  - MorphoSys Research Site, Tampere
- France (2):
  - MorphoSys Research Site, Grenoble
  - MorphoSys Research Site, Le Mans
- Germany (13):
  - MorphoSys Research Site, Aachen
  - MorphoSys Research Site, Berlin
  - MorphoSys Research Site, Düsseldorf
  - MorphoSys Research Site, Giessen
  - Morphosys Research Site, Homburg
  - MorphoSys Research Site, Leipzig
  - MorphoSys Research Site, Mainz
  - MorphoSys Research Site, Munich
  - MorphoSys Research Site, Mutlangen
  - Morphosys Research Site, Münster
  - MorphoSys Research Site, Rostock
  - MorphoSys Research Site, Stuttgart
  - MorphoSys, Traunstein
- Hungary (4):
  - MorphoSys, Budapest
  - MorphoSys Research Site, Debrecen
  - MorphoSys Research Site, Győr
  - MorphoSys, Szeged
- Israel (4):
  - MorphoSys Research Site, Haifa
  - MorphoSys Research Site, Jerusalem
  - MorphoSys Research Site, Kfar Saba
  - MorphoSys Research Site, Tel Aviv
- Italy (21):
  - MorphoSys Research Site, Alessandria
  - MorphoSys Research Site, Bologna
  - MorphoSys Research Site, Campobasso
  - MorphoSys Research Site, Cona
  - MorphoSys Research Site, Genova
  - MorphoSys Research Site, Lecce
  - MorphoSys Research Site, Meldola
  - MorphoSys Research Site, Monza
  - MorphoSys Research Site, Napoli
  - Morphosys Research Site, Novara
  - MorphoSys Research Site, Orbassano
  - MorphoSys Research Site, Parma
  - MorphoSys Research Site, Pavia
  - MorphoSys Research Site, Pisa
  - MorphoSys Research Site, Ravenna
  - MorphoSys Research Site, Reggio Emilia
  - MorphoSys Research Site, Rimini
  - MorphoSys Research Site, Rome
  - Morphosys Research Site, Terni
  - MorphoSys Research Site, Turin
  - Morphosys Research Site, Turin
- New Zealand (3):
  - MorphoSys Research Site, Addington
  - MorphoSys Research Site, Auckland
  - MorphoSys Research Site, Grafton
- Poland (8):
  - Morphosys Research Site, Bydgoszcz
  - MorphoSys Research Site, Gdynia
  - MorphoSys Research Site, Krakow
  - MorphoSys Research Site, Legnica
  - MorphoSys Research Site, Lodz
  - MorphoSys Research Site, Lublin
  - Morphosys Research Site, Warsaw
  - MorphoSys Research Site, Wroclaw
- Portugal (5):
  - MorphoSys Research Site, Braga
  - MorphoSys Research Site, Coimbra
  - MorphoSys Research Site, Matosinhos Municipality
  - MorphoSys Research Site, Porto
  - MorphoSys Research Site, Pragal
- Romania (2):
  - MorphoSys Research Site, Bucharest
  - MorphoSys Research Site, Iași
- Serbia (2):
  - MorphoSys Research Site, Belgrade
  - MorphoSys Research Site, Kragujevac
- MorphoSys Research Site, Singapore, Singapore
- South Korea (7):
  - MorphoSys Research Site, Busan
  - MorphoSys Research Site, Goyang-si
  - MorphoSys Research Site, Incheon
  - MorphoSys Research Site, Jeonju
  - MorphoSys Research Site, Seongnam
  - MorphoSys Research Site, Seoul
  - MorphoSys Research Site, Ulsan
- Spain (10):
  - MorphoSys Research Site, Cadiz
  - MorphoSys Research Site, Girona
  - MorphoSys Research Site, L'Hospitalet de Llobregat
  - MorphoSys Research Site, Madrid
  - MorphoSys Research Site, Palma de Mallorca
  - MorphoSys Research Site, Pamplona
  - MorphoSys Research Site, Pozuelo de Alarcón
  - MorphoSys, Sabadell
  - MorphoSys Research Site, Salamanca
  - MorphoSys Research Site, Valencia
- Taiwan (3):
  - Morphosys Research Site, Chang-hua
  - Morphosys Research Site, Hualien City
  - Morphosys Research Site, Taichung
- Turkey (Türkiye) (7):
  - MorphoSys Research Site, Adana
  - MorphoSys Research Site, Ankara
  - MorphoSys Research Site, Bornova
  - MorphoSys Research Site, Gaziantep
  - MorphoSys Research Site, Izmir
  - MorphoSys Research Site, Manisa
  - MorphoSys Research Site, Samsun
- United Kingdom (3):
  - Morphosys Research Site, Birmingham
  - MorphoSys Research Site, Leeds
  - MorphoSys Research Site, Southend-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 138 study centers in: Australia, Austria, Canada, Croatia, Czech Republic, Finland, France, Germany, Hungary, Israel, Italy, New Zealand, Poland, Portugal, Romania, Serbia, South Korea, Spain, Singapore, Taiwan, Turkey, the United Kingdom, and the United States of America.
Groups:
- Tafasitamab + Bendamustine: Participants received intravenous (IV) tafasitamab 12.0 milligrams per kilogram (mg/kg) in combination with IV bendamustine 90 mg/meters squared (m^2) in 28-day cycles for a maximum of 6 cycles. During Cycles 1 to 3, participants received tafastiamab on Days 1, 8, 15, and 22, plus a loading dose on Day 4 of Cycle 1. Participants received bendamustine on either Days 2 and 3 or Days 1 and 2 of Cycles 1 to 6. Participants with an ongoing response of at least partial response at the end of Cycle 6, as per local assessment, continued tafasitamab or rituximab monotherapy per initially allocated treatment until disease progression. Treatment was stopped due to disease progression, unacceptable toxicity, death, or discontinuation for any other reason, whichever came first.
- Rituximab + Bendamustine: Participants received IV rituximab 375 mg/m^2 in combination with IV bendamustine 90 mg/m^2 in 28-day cycles for a maximum of 6 cycles. Participants received rituximab on Day 1 of each cycle until disease progression. Participants received bendamustine on either Days 2 and 3 or Days 1 and 2 of Cycles 1 to 6. Participants with an ongoing response of at least partial response at the end of Cycle 6, as per local assessment, continued tafasitamab or rituximab monotherapy per initially allocated treatment until disease progression. Treatment was stopped due to disease progression, unacceptable toxicity, death, or discontinuation for any other reason, whichever came first.
Period: Overall Study
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Started | 226 | 227
Completed | 0 | 0
Not Completed | 226 | 227
Not completed — Adverse Event | 12 | 3
Not completed — Death | 123 | 123
Not completed — Lost to Follow-up | 6 | 7
Not completed — Noncompliance with Study Drug | 2 | 0
Not completed — Captured as "Other" in Database | 29 | 34
Not completed — Physician Decision | 1 | 7
Not completed — Progressive Disease | 24 | 27
Not completed — Completed the Maximum per Protocol Treatment Period | 1 | 0
Not completed — Diagnosed with COVID-19 and/or Tested Positive for Coronavirus SARS-CoV-2 | 2 | 1
Not completed — Withdrawal by Subject | 26 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine | Total
Number analyzed (Participants) | 226 | 227 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (10.36) | 70.8 (9.92) | 70.9 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 96 | 192
  Male | 130 | 131 | 261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian | 41 | 45 | 86
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 172 | 171 | 343
  Not Applicable in Enrolled Country | 8 | 4 | 12
  Captured as "Other" in Database | 2 | 2 | 4
  Iraqi | 1 | 0 | 1
  European | 0 | 2 | 2
  Eurasian | 0 | 1 | 1
  Captured as "Hispanic" in Database | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Progression-Free Survival by Independent Radiology/Clinical Review Committee Assessment in the Overall Population
Description: Progression-free survival was defined as the time from randomization to tumor progression or death from any cause.
Time Frame: up to 41.4 months
Population: Full Analysis Set (FAS): all participants who were randomized to either treatment arm. Participants were analyzed according to the treatment and stratification factors they were assigned to during the randomization procedure. 95% confidence intervals (CIs) (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
months | 7.10 [5.800 to 8.500] | 8.30 [5.600 to 11.500]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; p = 0.468, Inverse normal test; The Inverse Normal method combines information (p-value) from the interim analysis and information from the final analysis; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.837 to 1.351] — The hazard ratio estimate for treatment was based on a stratified Cox model with stratification factors as per the Interactive Web Response System (IWRS). Rituximab + bendamustine was the reference treatment group

2. Primary Outcome: Kaplan-Meier Estimate of Progression-Free Survival by Independent Radiology/Clinical Review Committee Assessment in the Natural Killer Cell Count-Low Subgroup
Description: Progression-free survival was defined as the time from randomization to tumor progression or death from any cause.
Time Frame: up to 46.5 months
Population: Natural Killer Cell Count-Low Full Analysis Set: participants in the FAS with ≤100 NK cells/µL at Baseline. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
months | 5.60 [4.400 to 8.600] | 5.60 [3.600 to 10.000]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; p = 0.568, Inverse normal test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.586 to 1.330] — The hazard ratio estimate for treatment was based on a stratified Cox model with stratification factors as per the Interactive Web Response System. Rituximab + bendamustine is the reference treatment group

3. Secondary Outcome: Best Objective Response Rate (ORR) by Independent Radiology/Clinical Review Committee Assessment in the Overall Population
Description: Best ORR was defined as the percentage of patients with complete response (CR) or partial response (PR) based on the best response achieved at any time during the study. Per International Working Group response criteria: CR: the disappearance of all evidence of disease; PR: regression of measurable disease and no new sites.
Time Frame: up to 77 months
Population: Full Analysis Set. A 2-sided 95% Clopper-Pearson exact method based on binomial distribution was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
percentage of participants | 65.5 [58.90 to 71.67] | 61.7 [55.01 to 68.03]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.812 to 1.779]; A Cochran-Mantel-Haenszel (CMH) test stratified by Baseline stratification factors was performed for response variable coded as follows: 1 for response (CR or PR) and 0 for nonresponse (stable disease [SD] or progressive disease [PD] or unknown)

4. Secondary Outcome: Best ORR by Independent Radiology/Clinical Review Committee Assessment in the Natural Killer Cell Count-Low Subgroup
Description: Best ORR was defined as the percentage of patients with CR or PR based on the best response achieved at any time during the study. Per International Working Group response criteria: CR: the disappearance of all evidence of disease; PR: regression of measurable disease and no new sites.
Time Frame: up to 77 months
Population: Natural Killer Cell Count-Low Full Analysis Set. A 2-sided 95% Clopper-Pearson exact method based on binomial distribution was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
percentage of participants | 64.8 [53.86 to 74.66] | 59.5 [47.41 to 70.73]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.778 to 3.041]; [other analysis details as in outcome 3, analysis 1]

5. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response by Independent Radiology/Clinical Review Committee Assessment in the Overall Population
Description: Duration of response was defined as the elapsed time (in months) between the date of the first documented response (CR or PR) and the following date of an event defined as the first documented progression (any new lesion or an increase by ≥50% of previously involved sites from nadir) or death. Per International Working Group response criteria: CR: the disappearance of all evidence of disease; PR: regression of measurable disease and no new sites.
Time Frame: up to 40.2 months
Population: Full Analysis Set. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley. Only participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 148 | 140
months | 7.40 [5.800 to 12.100] | 12.10 [10.000 to 23.300]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.938 to 1.745]; The hazard ratio estimate for treatment was based on a stratified Cox model with stratification factors as per IWRS. Rituximab + bendamustine was the reference treatment group

6. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response by Independent Radiology/Clinical Review Committee Assessment in the Natural Killer Cell Count-Low Subgroup
Description: as for outcome 5
Time Frame: up to 44.7 months
Population: Natural Killer Cell Count-Low Full Analysis Set. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley. Only participants with CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 57 | 44
months | 6.70 [3.700 to 12.700] | 10.30 [4.900 to 37.500]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.673 to 2.035]; [other analysis details as in outcome 5, analysis 1]

7. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival in the Overall Population
Description: Overall survival was defined as the time (in months) from randomization until death from any cause.
Time Frame: up to 50.0 months
Population: Full Analysis Set. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
months | 14.60 [11.600 to 23.400] | 20.20 [13.400 to 24.300]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.875 to 1.452]; [other analysis details as in outcome 5, analysis 1]

8. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival in the Natural Killer Cell Count-Low Subgroup
Description: Overall survival was defined as the time (in months) from randomization until death from any cause.
Time Frame: up to 50.6 months
Population: Natural Killer Cell Count-Low Full Analysis Set. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
months | 10.60 [8.300 to 19.700] | 12.50 [8.300 to 32.300]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.682 to 1.626]; [other analysis details as in outcome 5, analysis 1]

9. Secondary Outcome: Disease Control Rate (DCR) by Independent Radiology/Clinical Review Committee Assessment in the Overall Population
Description: DCR was defined as the percentage of participants with a CR, PR, or stable disease (SD) based on the best response achieved at any time during the study. Per the International Working Group response criteria: CR: the disappearance of all evidence of disease; PR: regression of measurable disease and no new sites; SD: failure to attain CR/PR or progressive disease (PD; any new lesion or an increase by ≥50% of previously involved sites from nadir).
Time Frame: up to 77 months
Population: Full Analysis Set. A 2-sided 95% Clopper-Pearson exact method based on binomial distribution was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
percentage of participants | 76.1 [70.00 to 81.51] | 71.8 [65.47 to 77.56]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.829 to 1.985]; A CMH test stratified by Baseline stratification factors was performed for response variable coded as follows: 1 for response (CR or PR) and 0 for nonresponse (stable disease [SD] or progressive disease [PD] or unknown)

10. Secondary Outcome: DCR by Independent Radiology/Clinical Review Committee Assessment in the Natural Killer Cell Count-Low Subgroup
Description: DCR was defined as the percentage of participants with a CR, PR, or SD based on the best response achieved at any time during the study. Per the International Working Group response criteria: CR: the disappearance of all evidence of disease; PR: regression of measurable disease and no new sites; SD: failure to attain CR/PR or PD (any new lesion or an increase by ≥50% of previously involved sites from nadir).
Time Frame: up to 77 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
percentage of participants | 75.0 [64.63 to 83.62] | 70.3 [58.52 to 80.34]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.755 to 3.457]; [other analysis details as in outcome 9, analysis 1]

11. Secondary Outcome: Kaplan-Meier Estimate of Time to Progression by Independent Radiology/Clinical Review Committee Assessment in the Overall Population
Description: Time to progression was defined as the time (in months) from randomization until documented diffuse large B-call lymphoma (DLBCL) progression or death as a result of lymphoma. Death from other causes than lymphoma was not considered in relation to the TTP evaluation.
Time Frame: up to 25.8 months
Population: Full Analysis Set. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley. Only participants with progression/death as a result of lymphoma were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 117 | 111
months | 8.20 [6.200 to 9.300] | 11.10 [8.100 to 18.300]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.831 to 1.416]; [other analysis details as in outcome 5, analysis 1]

12. Secondary Outcome: Kaplan-Meier Estimate of Time to Progression by Independent Radiology/Clinical Review Committee Assessment in the Natural Killer Cell Count-Low Subgroup
Description: as for outcome 11
Time Frame: up to 40.6 months
Population: Natural Killer Cell Count-Low Full Analysis Set. 95% CIs (Greenwood formula) for the median and the 25th and 75th percentiles were calculated using the method of Brookmeyer and Crowley. Only participants with progression/death as a result of lymphoma were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 50 | 36
months | 8.00 [5.400 to 9.200] | 10.00 [3.800 to 39.400]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.633 to 1.595]; [other analysis details as in outcome 5, analysis 1]

13. Secondary Outcome: Kaplan-Meier Estimate of Time to Next Treatment in the Overall Population
Description: Time to next treatment was defined as the time (in months) from randomization to the institution of the next anti-neoplastic therapy (for any reason including disease progression, treatment toxicity, and participant preference) or death due to any cause, whatever came first.
Time Frame: up to 59.4 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
months | 8.80 [7.500 to 10.900] | 8.70 [6.800 to 11.500]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.794 to 1.244]; [other analysis details as in outcome 5, analysis 1]

14. Secondary Outcome: Kaplan-Meier Estimate of Time to Next Treatment in the Natural Killer Cell Count-Low Subgroup
Description: as for outcome 13
Time Frame: up to 70.1 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
months | 7.20 [5.800 to 9.500] | 6.30 [4.300 to 9.000]
Statistical Analysis 1: Comparison: Tafasitamab + Bendamustine vs Rituximab + Bendamustine; Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.570 to 1.220]; [other analysis details as in outcome 5, analysis 1]

15. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event was defined as any untoward medical occurrence in a participant administered a medicinal product, which did not necessarily have a causal relationship to this treatment. An AE could therefore have been any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it was considered related to that study drug. TEAEs were defined as any adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: up to 77 months
Population: Safety Analysis Set: all participants who received at least one dose of tafasitamab, bendamustine, or rituximab. Analyses were based on the actual treatment received.
Measure: Number; unit: participants
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 219 | 225
participants | 215 | 215

16. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE
Description: AEs were graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 (or higher). Grade 1: mild; asymptomatic or mild symptoms. Grade 2: moderate. Grade 3: severe or medically significant but not immediately life threatening. Grade 4: life-threatening consequences. Grade 5: death. TEAEs were defined as any adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: up to 77 months
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 219 | 225
participants | 191 | 159

17. Secondary Outcome: Change From Baseline (CFB) in the EORTC QLQ-C30 Scores at End of Treatment in the Overall Population
Description: The European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) contains 30 items and measures 5 functional dimensions (i.e., physical, role, emotional, cognitive, and social), 3 symptom items (i.e., fatigue, nausea/vomiting, and pain), 6 single items (i.e., dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and financial impact), and a global health and quality of life scale. For each scale and single item, a linear transformation was applied to standardize the scores between 0 (worst) and 100 (best) as described in the EORTC QLQ-C30 Scoring Manual.
Time Frame: Baseline; End of Treatment (EOT) (up to 77 months)
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
scores on a scale
  Baseline; Global Health Status/QoL Scale: number analyzed (Participants) | 223 | 225
  Baseline; Global Health Status/QoL Scale | 59.19 (22.94) | 59.89 (23.75)
  Baseline; Physical Functioning: number analyzed (Participants) | 222 | 225
  Baseline; Physical Functioning | 71.68 (23.05) | 69.39 (24.60)
  Baseline; Role Functioning: number analyzed (Participants) | 221 | 226
  Baseline; Role Functioning | 68.91 (30.84) | 69.53 (31.48)
  Baseline; Emotional Functioning: number analyzed (Participants) | 220 | 224
  Baseline; Emotional Functioning | 76.63 (22.24) | 74.79 (25.05)
  Baseline; Cognitive Functioning: number analyzed (Participants) | 222 | 224
  Baseline; Cognitive Functioning | 82.81 (18.61) | 81.41 (22.74)
  Baseline; Social Functioning: number analyzed (Participants) | 222 | 224
  Baseline; Social Functioning | 74.74 (27.53) | 73.93 (29.45)
  Baseline, Fatigue: number analyzed (Participants) | 221 | 223
  Baseline, Fatigue | 37.74 (26.69) | 36.64 (27.28)
  Baseline, Nausea and Vomiting: number analyzed (Participants) | 222 | 225
  Baseline, Nausea and Vomiting | 6.20 (15.26) | 9.69 (21.25)
  Baseline, Pain: number analyzed (Participants) | 220 | 223
  Baseline, Pain | 28.25 (31.02) | 27.36 (30.18)
  Baseline, Dyspnoea: number analyzed (Participants) | 223 | 227
  Baseline, Dyspnoea | 19.43 (25.13) | 18.06 (25.70)
  Baseline, Insomnia: number analyzed (Participants) | 223 | 227
  Baseline, Insomnia | 30.64 (32.77) | 29.22 (31.87)
  Baseline, Loss of Appetite: number analyzed (Participants) | 222 | 227
  Baseline, Loss of Appetite | 20.27 (28.44) | 22.17 (31.87)
  Baseline, Constipation: number analyzed (Participants) | 223 | 227
  Baseline, Constipation | 15.25 (24.85) | 14.83 (24.30)
  Baseline, Diarrhoea: number analyzed (Participants) | 223 | 225
  Baseline, Diarrhoea | 8.07 (17.46) | 8.74 (21.07)
  Baseline, Financial Impact: number analyzed (Participants) | 223 | 225
  Baseline, Financial Impact | 14.20 (24.97) | 21.78 (28.26)
  CFB at EOT; Baseline; Global Health Status/QoL Scale: number analyzed (Participants) | 128 | 145
  CFB at EOT; Baseline; Global Health Status/QoL Scale | -7.23 (22.56) | -7.99 (22.71)
  CFB at EOT; Baseline; Physical Functioning: number analyzed (Participants) | 128 | 144
  CFB at EOT; Baseline; Physical Functioning | -13.59 (25.48) | -7.51 (22.95)
  CFB at EOT; Role Functioning: number analyzed (Participants) | 128 | 144
  CFB at EOT; Role Functioning | -14.84 (33.87) | -10.88 (32.35)
  CFB at EOT; Emotional Functioning: number analyzed (Participants) | 128 | 144
  CFB at EOT; Emotional Functioning | -5.60 (24.88) | -2.41 (24.83)
  CFB at EOT; Cognitive Functioning: number analyzed (Participants) | 128 | 145
  CFB at EOT; Cognitive Functioning | -7.29 (23.37) | -4.71 (24.67)
  CFB at EOT; Social Functioning: number analyzed (Participants) | 128 | 144
  CFB at EOT; Social Functioning | -14.32 (31.56) | -4.98 (27.03)
  CFB at EOT, Fatigue: number analyzed (Participants) | 128 | 146
  CFB at EOT, Fatigue | 11.89 (31.49) | 10.24 (24.30)
  CFB at EOT, Nausea and Vomiting: number analyzed (Participants) | 128 | 145
  CFB at EOT, Nausea and Vomiting | 5.47 (18.37) | 3.10 (25.00)
  CFB at EOT, Pain: number analyzed (Participants) | 129 | 145
  CFB at EOT, Pain | 6.33 (30.42) | 7.93 (33.11)
  CFB at EOT, Dyspnoea: number analyzed (Participants) | 128 | 145
  CFB at EOT, Dyspnoea | 9.11 (34.93) | 8.05 (28.40)
  CFB at EOT, Insomnia: number analyzed (Participants) | 128 | 146
  CFB at EOT, Insomnia | 1.30 (36.80) | 2.28 (33.37)
  CFB at EOT, Loss of Appetite: number analyzed (Participants) | 128 | 146
  CFB at EOT, Loss of Appetite | 16.15 (38.33) | 9.36 (31.98)
  CFB at EOT, Constipation: number analyzed (Participants) | 128 | 146
  CFB at EOT, Constipation | 5.21 (33.58) | 1.60 (28.05)
  CFB at EOT, Diarrhoea: number analyzed (Participants) | 128 | 145
  CFB at EOT, Diarrhoea | 7.03 (28.26) | 1.38 (28.02)
  CFB at EOT, Financial Impact: number analyzed (Participants) | 128 | 142
  CFB at EOT, Financial Impact | 2.08 (22.04) | 1.17 (25.24)

18. Secondary Outcome: Change From Baseline (CFB) in the EORTC QLQ-C30 Scores at End of Treatment in the Natural Killer Cell Count-Low Subgroup
Description: as for outcome 17
Time Frame: Baseline; End of Treatment (EOT) (up to 77 months)
Population: Natural Killer Cell Count-Low Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
scores on a scale
  Baseline; Global Health Status/QoL Scale: number analyzed (Participants) | 86 | 74
  Baseline; Global Health Status/QoL Scale | 57.66 (22.37) | 52.59 (24.13)
  Baseline; Physical Functioning: number analyzed (Participants) | 86 | 72
  Baseline; Physical Functioning | 68.60 (24.73) | 64.30 (26.46)
  Baseline; Role Functioning: number analyzed (Participants) | 85 | 74
  Baseline; Role Functioning | 65.89 (31.61) | 60.59 (33.63)
  Baseline; Emotional Functioning: number analyzed (Participants) | 85 | 73
  Baseline; Emotional Functioning | 76.10 (22.32) | 67.61 (28.71)
  Baseline; Cognitive Functioning: number analyzed (Participants) | 86 | 74
  Baseline; Cognitive Functioning | 84.88 (18.72) | 77.03 (23.84)
  Baseline; Social Functioning: number analyzed (Participants) | 86 | 73
  Baseline; Social Functioning | 73.84 (27.00) | 67.34 (31.87)
  Baseline, Fatigue: number analyzed (Participants) | 85 | 72
  Baseline, Fatigue | 39.02 (26.61) | 43.62 (28.01)
  Baseline, Nausea and Vomiting: number analyzed (Participants) | 86 | 74
  Baseline, Nausea and Vomiting | 6.20 (14.24) | 15.77 (26.44)
  Baseline, Pain: number analyzed (Participants) | 85 | 72
  Baseline, Pain | 28.88 (32.38) | 34.68 (32.50)
  Baseline, Dyspnoea: number analyzed (Participants) | 86 | 74
  Baseline, Dyspnoea | 21.32 (25.52) | 21.62 (28.37)
  Baseline, Insomnia: number analyzed (Participants) | 86 | 74
  Baseline, Insomnia | 31.78 (30.64) | 36.49 (33.64)
  Baseline, Loss of Appetite: number analyzed (Participants) | 86 | 74
  Baseline, Loss of Appetite | 21.32 (27.49) | 29.73 (36.00)
  Baseline, Constipation: number analyzed (Participants) | 86 | 74
  Baseline, Constipation | 17.83 (26.91) | 16.67 (27.72)
  Baseline, Diarrhoea: number analyzed (Participants) | 86 | 74
  Baseline, Diarrhoea | 7.75 (16.71) | 9.01 (22.95)
  Baseline, Financial Impact: number analyzed (Participants) | 86 | 74
  Baseline, Financial Impact | 13.57 (25.25) | 24.32 (32.78)
  CFB at EOT; Baseline; Global Health Status/QoL Scale: number analyzed (Participants) | 52 | 42
  CFB at EOT; Baseline; Global Health Status/QoL Scale | -6.57 (23.70) | -7.54 (30.84)
  CFB at EOT; Baseline; Physical Functioning: number analyzed (Participants) | 51 | 41
  CFB at EOT; Baseline; Physical Functioning | -15.29 (25.83) | -11.83 (33.60)
  CFB at EOT; Role Functioning: number analyzed (Participants) | 51 | 41
  CFB at EOT; Role Functioning | -19.61 (37.07) | -15.45 (41.06)
  CFB at EOT; Emotional Functioning: number analyzed (Participants) | 52 | 41
  CFB at EOT; Emotional Functioning | -4.81 (28.02) | 0.27 (33.98)
  CFB at EOT; Cognitive Functioning: number analyzed (Participants) | 52 | 42
  CFB at EOT; Cognitive Functioning | -7.69 (22.01) | -5.95 (30.54)
  CFB at EOT; Social Functioning: number analyzed (Participants) | 52 | 41
  CFB at EOT; Social Functioning | -16.67 (27.42) | -2.44 (32.18)
  CFB at EOT, Fatigue: number analyzed (Participants) | 51 | 42
  CFB at EOT, Fatigue | 13.51 (31.69) | 13.10 (33.19)
  CFB at EOT, Nausea and Vomiting: number analyzed (Participants) | 51 | 41
  CFB at EOT, Nausea and Vomiting | 5.66 (14.78) | -3.66 (34.86)
  CFB at EOT, Pain: number analyzed (Participants) | 52 | 42
  CFB at EOT, Pain | 8.65 (33.09) | 7.94 (42.97)
  CFB at EOT, Dyspnoea: number analyzed (Participants) | 51 | 42
  CFB at EOT, Dyspnoea | 9.15 (37.17) | 7.94 (32.77)
  CFB at EOT, Insomnia: number analyzed (Participants) | 51 | 42
  CFB at EOT, Insomnia | 5.88 (35.09) | -1.59 (41.62)
  CFB at EOT, Loss of Appetite: number analyzed (Participants) | 51 | 42
  CFB at EOT, Loss of Appetite | 20.26 (41.14) | 10.32 (42.60)
  CFB at EOT, Constipation: number analyzed (Participants) | 51 | 42
  CFB at EOT, Constipation | 5.88 (32.46) | 0.79 (30.79)
  CFB at EOT, Diarrhoea: number analyzed (Participants) | 52 | 42
  CFB at EOT, Diarrhoea | 5.77 (21.61) | 5.56 (30.28)
  CFB at EOT, Financial Impact: number analyzed (Participants) | 52 | 41
  CFB at EOT, Financial Impact | 2.56 (17.27) | 7.32 (26.37)

19. Secondary Outcome: Change From Baseline (CFB) in EQ-5D-5L Dimension Scores at End of Treatment in the Overall Population
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome. The EQ-5D-5L descriptive system is composed of 5 dimensions (mobility, self-case, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 response levels, which are coded by single-digit numbers: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems, 5 = unable to/extreme problems. The EQ-5D-5L also includes a graded (0 [worst overall health] to 100 [best overall health]) vertical visual analog scale that provides a quantitative measure of the participant's perception of their overall health.
Time Frame: Baseline; End of Treatment (EOT) (up to 77 months)
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
scores on a scale
  Baseline, Mobility Level: number analyzed (Participants) | 206 | 212
  Baseline, Mobility Level | 1.83 (0.969) | 1.94 (1.054)
  Baseline, Self-care Level: number analyzed (Participants) | 206 | 212
  Baseline, Self-care Level | 1.37 (0.771) | 1.44 (0.861)
  Baseline, Usual Activities: number analyzed (Participants) | 206 | 212
  Baseline, Usual Activities | 1.97 (1.086) | 1.92 (1.063)
  Baseline, Pain/Discomfort: number analyzed (Participants) | 206 | 211
  Baseline, Pain/Discomfort | 2.04 (1.045) | 2.08 (1.027)
  Baseline, Anxiety/Depression: number analyzed (Participants) | 206 | 212
  Baseline, Anxiety/Depression | 1.67 (0.844) | 1.73 (0.907)
  CFB at EOT, Mobility Level: number analyzed (Participants) | 118 | 132
  CFB at EOT, Mobility Level | 0.47 (1.076) | 0.25 (1.094)
  CFB at EOT, Self-care Level: number analyzed (Participants) | 118 | 132
  CFB at EOT, Self-care Level | 0.48 (1.052) | 0.23 (0.946)
  CFB at EOT, Usual Activities: number analyzed (Participants) | 118 | 131
  CFB at EOT, Usual Activities | 0.42 (1.410) | 0.31 (1.066)
  CFB at EOT, Pain/Discomfort: number analyzed (Participants) | 118 | 131
  CFB at EOT, Pain/Discomfort | 0.29 (1.102) | 0.09 (1.173)
  CFB at EOT, Anxiety/Depression: number analyzed (Participants) | 118 | 131
  CFB at EOT, Anxiety/Depression | 0.33 (1.071) | 0.21 (1.030)

20. Secondary Outcome: Change From Baseline (CFB) in EQ-5D-5L VAS Score at End of Treatment in the Overall Population
Description: as for outcome 19
Time Frame: Baseline; End of Treatment (EOT) (up to 77 months)
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 226 | 227
scores on a scale
  Baseline: number analyzed (Participants) | 206 | 211
  Baseline | 66.22 (20.5) | 66.69 (20.4)
  Change from Baseline at End of Treatment: number analyzed (Participants) | 119 | 129
  Change from Baseline at End of Treatment | -8.10 (21.1) | -5.47 (23.2)

21. Secondary Outcome: Change From Baseline (CFB) in EQ-5D-5L VAS Score at End of Treatment in the Natural Killer Cell Count-Low Subgroup
Description: as for outcome 19
Time Frame: Baseline; End of Treatment (EOT) (up to 77 months)
Population: Natural Killer Cell Count-Low Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
scores on a scale
  Baseline: number analyzed (Participants) | 78 | 68
  Baseline | 65.87 (21.4) | 58.65 (20.7)
  Change from Baseline at End of Treatment: number analyzed (Participants) | 48 | 38
  Change from Baseline at End of Treatment | -10.75 (21.0) | -7.53 (31.4)

22. Secondary Outcome: Change From Baseline (CFB) in EQ-5D-5L Dimension Scores at End of Treatment in the Natural Killer Cell Count-Low Subgroup
Description: as for outcome 19
Time Frame: Baseline; End of Treatment (EOT) (up to 77 months)
Population: Natural Killer Cell Count-Low Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 88 | 74
scores on a scale
  Baseline, Mobility Level: number analyzed (Participants) | 78 | 69
  Baseline, Mobility Level | 2.09 (0.983) | 2.04 (1.104)
  Baseline, Self-care Level: number analyzed (Participants) | 78 | 69
  Baseline, Self-care Level | 1.49 (0.977) | 1.54 (0.917)
  Baseline, Usual Activities: number analyzed (Participants) | 78 | 69
  Baseline, Usual Activities | 2.03 (1.116) | 2.14 (1.228)
  Baseline, Pain/Discomfort: number analyzed (Participants) | 78 | 68
  Baseline, Pain/Discomfort | 2.08 (1.054) | 2.26 (1.060)
  Baseline, Anxiety/Depression: number analyzed (Participants) | 78 | 69
  Baseline, Anxiety/Depression | 1.65 (0.803) | 1.96 (1.143)
  CFB at EOT, Mobility Level: number analyzed (Participants) | 47 | 39
  CFB at EOT, Mobility Level | 0.55 (1.080) | 0.46 (1.315)
  CFB at EOT, Self-care Level: number analyzed (Participants) | 47 | 39
  CFB at EOT, Self-care Level | 0.53 (1.080) | 0.41 (1.312)
  CFB at EOT, Usual Activities: number analyzed (Participants) | 47 | 38
  CFB at EOT, Usual Activities | 0.62 (1.392) | 0.53 (1.224)
  CFB at EOT, Pain/Discomfort: number analyzed (Participants) | 47 | 38
  CFB at EOT, Pain/Discomfort | 0.40 (1.173) | 0.05 (1.469)
  CFB at EOT, Anxiety/Depression: number analyzed (Participants) | 47 | 38
  CFB at EOT, Anxiety/Depression | 0.30 (1.250) | 0.24 (1.324)

23. Secondary Outcome: Tafasitamab Serum Concentrations
Description: Blood samples were collected for the assessment of serum concentrations of tafasitamab.
Time Frame: pre-dose: Cycle 1 Days 1, 2, 3, 4, 15; Cycle 2 Days 1, 15; Cycle 3 Days 1, 15, Cycles 4, 5, 6, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, and 35 Day 1. 1 hour post-dose: Cycle 1 Days 1, 4, 15; Cycle 2 Days 1, 15; Cycle 3 Days 1, 15
Population: Pharmacokinetic (PK) Analysis Set: all participants who received at least one dose of tafasitamab and had at least one quantifiable serum tafasitamab concentration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
Number analyzed (Participants) | 219 | 0
micrograms per milliliter (µg/mL)
  Cycle 1 Day 1, pre-dose: number analyzed (Participants) | 218 | 0
  Cycle 1 Day 1, pre-dose | 0.00 (58.8) |
  Cycle 1 Day 1, 1 hour post-dose: number analyzed (Participants) | 40 | 0
  Cycle 1 Day 1, 1 hour post-dose | 2.45 (37.1) |
  Cycle 1 Day 2, pre-dose: number analyzed (Participants) | 215 | 0
  Cycle 1 Day 2, pre-dose | 2.06 (30.2) |
  Cycle 1 Day 3, pre-dose: number analyzed (Participants) | 211 | 0
  Cycle 1 Day 3, pre-dose | 1.63 (30.4) |
  Cycle 1 Day 4, pre-dose: number analyzed (Participants) | 209 | 0
  Cycle 1 Day 4, pre-dose | 1.34 (33.5) |
  Cycle 1 Day 4, 1 hour post-dose: number analyzed (Participants) | 169 | 0
  Cycle 1 Day 4, 1 hour post-dose | 3.84 (31.8) |
  Cycle 1 Day 15, pre-dose: number analyzed (Participants) | 198 | 0
  Cycle 1 Day 15, pre-dose | 2.14 (39.1) |
  Cycle 1 Day 15, 1 hour post-dose: number analyzed (Participants) | 168 | 0
  Cycle 1 Day 15, 1 hour post-dose | 4.68 (31.9) |
  Cycle 2 Day 1, pre-dose: number analyzed (Participants) | 197 | 0
  Cycle 2 Day 1, pre-dose | 2.37 (55.1) |
  Cycle 2 Day 1, 1 hour post-dose: number analyzed (Participants) | 160 | 0
  Cycle 2 Day 1, 1 hour post-dose | 4.80 (32.8) |
  Cycle 2 Day 15, pre-dose: number analyzed (Participants) | 174 | 0
  Cycle 2 Day 15, pre-dose | 2.73 (42.4) |
  Cycle 2 Day 15, 1 hour post-dose: number analyzed (Participants) | 152 | 0
  Cycle 2 Day 15, 1 hour post-dose | 5.20 (44.4) |
  Cycle 3 Day 1, pre-dose: number analyzed (Participants) | 174 | 0
  Cycle 3 Day 1, pre-dose | 2.92 (43.5) |
  Cycle 3 Day 1, 1 hour post-dose: number analyzed (Participants) | 134 | 0
  Cycle 3 Day 1, 1 hour post-dose | 5.38 (32.2) |
  Cycle 3 Day 15, pre-dose: number analyzed (Participants) | 159 | 0
  Cycle 3 Day 15, pre-dose | 3.14 (38.3) |
  Cycle 3 Day 15, 1 hour post-dose: number analyzed (Participants) | 136 | 0
  Cycle 3 Day 15, 1 hour post-dose | 5.54 (30.1) |
  Cycle 4 Day 1, pre-dose: number analyzed (Participants) | 150 | 0
  Cycle 4 Day 1, pre-dose | 3.27 (43.2) |
  Cycle 5 Day 1, pre-dose: number analyzed (Participants) | 133 | 0
  Cycle 5 Day 1, pre-dose | 1.95 (54.6) |
  Cycle 6 Day 1, pre-dose: number analyzed (Participants) | 118 | 0
  Cycle 6 Day 1, pre-dose | 1.60 (61.2) |
  Cycle 7 Day 1, pre-dose: number analyzed (Participants) | 91 | 0
  Cycle 7 Day 1, pre-dose | 1.14 (75.3) |
  Cycle 9 Day 1, pre-dose: number analyzed (Participants) | 66 | 0
  Cycle 9 Day 1, pre-dose | 1.79 (50.3) |
  Cycle 11 Day 1, pre-dose: number analyzed (Participants) | 50 | 0
  Cycle 11 Day 1, pre-dose | 1.73 (58.1) |
  Cycle 13 Day 1, pre-dose: number analyzed (Participants) | 46 | 0
  Cycle 13 Day 1, pre-dose | 1.81 (66.4) |
  Cycle 15 Day 1, pre-dose: number analyzed (Participants) | 39 | 0
  Cycle 15 Day 1, pre-dose | 1.83 (55.8) |
  Cycle 17 Day 1, pre-dose: number analyzed (Participants) | 33 | 0
  Cycle 17 Day 1, pre-dose | 1.86 (48.3) |
  Cycle 19 Day 1, pre-dose: number analyzed (Participants) | 30 | 0
  Cycle 19 Day 1, pre-dose | 1.98 (36.4) |
  Cycle 21 Day 1, pre-dose: number analyzed (Participants) | 32 | 0
  Cycle 21 Day 1, pre-dose | 1.91 (52.0) |
  Cycle 23 Day 1, pre-dose: number analyzed (Participants) | 31 | 0
  Cycle 23 Day 1, pre-dose | 1.88 (55.2) |
  Cycle 25 Day 1, pre-dose: number analyzed (Participants) | 7 | 0
  Cycle 25 Day 1, pre-dose | 2.24 (37.7) |
  Cycle 27 Day 1, pre-dose: number analyzed (Participants) | 2 | 0
  Cycle 27 Day 1, pre-dose | 1.92 (12.6) |
  Cycle 29 Day 1, pre-dose: number analyzed (Participants) | 2 | 0
  Cycle 29 Day 1, pre-dose | 2.05 (21.3) |
  Cycle 31 Day 1, pre-dose: number analyzed (Participants) | 2 | 0
  Cycle 31 Day 1, pre-dose | 1.64 (23.9) |
  Cycle 33 Day 1, pre-dose: number analyzed (Participants) | 1 | 0
  Cycle 33 Day 1, pre-dose | 1.45 (NA) — Dispersion cannot be calculated for a single participant. |
  Cycle 35 Day 1, pre-dose: number analyzed (Participants) | 2 | 0
  Cycle 35 Day 1, pre-dose | 1.51 (2.7) |

ADVERSE EVENTS:
Time Frame: up to approximately 7.5 years
Description: All-Cause Mortality was assessed in the Full Analysis Set, comprised of all participants who were randomized to either treatment arm. Adverse events have been reported for the Safety Analysis Set, comprised of all participants who received at least one dose of tafasitamab, bendamustine, or rituximab.
Arm/Group | Tafasitamab + Bendamustine | Rituximab + Bendamustine
All-Cause Mortality (participants affected / at risk) | 129/226 | 127/227
Serious Adverse Events (participants affected / at risk) | 115/219 | 100/225
Other Adverse Events (participants affected / at risk) | 206/219 | 199/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafasitamab + Bendamustine (N=219) | Rituximab + Bendamustine (N=225)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (3)
COVID-19 (Infections and infestations) | 9 (9) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 6 (6)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (2)
Clostridial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulum oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 6 (7)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flatback syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Haemophilus sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 4 (4) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster reactivation (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Illness (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (3) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 5 (5)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Limbic encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Neutropenic sepsis (Infections and infestations) | 3 (3) | 0 (0)
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 26 (29) | 17 (17)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 9 (12) | 5 (5)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 4 (4)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (2) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (3)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Weil's disease (Infections and infestations) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tafasitamab + Bendamustine (N=219) | Rituximab + Bendamustine (N=225)
Abdominal pain (Gastrointestinal disorders) | 31 (41) | 15 (16)
Alanine aminotransferase increased (Investigations) | 11 (14) | 10 (16)
Anaemia (Blood and lymphatic system disorders) | 60 (94) | 48 (73)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (19) | 11 (11)
Aspartate aminotransferase increased (Investigations) | 12 (15) | 8 (13)
Asthenia (General disorders) | 40 (51) | 25 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (19) | 26 (30)
Blood creatinine increased (Investigations) | 18 (25) | 10 (17)
Constipation (Gastrointestinal disorders) | 50 (63) | 41 (46)
Cough (Respiratory, thoracic and mediastinal disorders) | 41 (68) | 25 (33)
Decreased appetite (Metabolism and nutrition disorders) | 47 (63) | 36 (45)
Diarrhoea (Gastrointestinal disorders) | 58 (103) | 43 (61)
Dizziness (Nervous system disorders) | 26 (32) | 14 (15)
Dyspepsia (Gastrointestinal disorders) | 18 (24) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (33) | 18 (21)
Fatigue (General disorders) | 56 (78) | 37 (45)
Headache (Nervous system disorders) | 30 (38) | 25 (36)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (31) | 15 (33)
Hypertension (Vascular disorders) | 13 (16) | 11 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 28 (48) | 30 (41)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (15) | 7 (10)
Hypotension (Vascular disorders) | 17 (18) | 12 (12)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (8) | 15 (15)
Insomnia (Psychiatric disorders) | 20 (22) | 18 (21)
Leukopenia (Blood and lymphatic system disorders) | 21 (37) | 14 (40)
Lymphopenia (Blood and lymphatic system disorders) | 20 (26) | 19 (39)
Nasopharyngitis (Infections and infestations) | 13 (15) | 14 (17)
Nausea (Gastrointestinal disorders) | 77 (133) | 62 (92)
Neutropenia (Blood and lymphatic system disorders) | 116 (304) | 98 (347)
Oedema peripheral (General disorders) | 25 (30) | 17 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (20) | 9 (10)
Pneumonia (Infections and infestations) | 9 (10) | 12 (13)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (18) | 26 (32)
Pyrexia (General disorders) | 38 (57) | 35 (49)
Rash (Skin and subcutaneous tissue disorders) | 18 (22) | 14 (18)
Tachycardia (Cardiac disorders) | 13 (14) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 67 (112) | 60 (101)
Upper respiratory tract infection (Infections and infestations) | 18 (29) | 21 (31)
Urinary tract infection (Infections and infestations) | 17 (21) | 20 (31)
Vomiting (Gastrointestinal disorders) | 31 (43) | 22 (38)
Weight decreased (Investigations) | 15 (15) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT02763319/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT02763319/SAP_001.pdf